CLINICAL TRIAL: NCT07102771
Title: The Efficacy of Hyaluronidase as an Adjuvant to Bupivacaine in Ultrasound-guided Erector Spinae Plane Block in Percutaneous Nephrolithotomy. Randomized Double-blind Controlled Study
Brief Title: Efficacy of Hyaluronidase Added to Bupivacaine in Ultrasound-guided Erector Spinae Plane Block in Percutaneous Nephrolithotomy.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Emad Mohamed Ahmed Abdelhafez, Lecturer of Anesthesia, Critical Care and Pain Management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-186-2025
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Erector Spinae Plane Block, Nephrolithotomy, Hyaluronidase

STUDY DESIGN:
Intervention Model Description: Controlled arm and interventional arm
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: ESPN with bupivacain 0.25% (Active Comparator): ESPN with (30 ml volume : 15 ml saline Plus 15 ml plain bupivacaine ) .
  Interventions: Procedure: Ultrasound guided erector spinae plane block
- Group II : ESPN with bupivacaine 0.25 % and hyalurinidase (Active Comparator): ESPN with ( 14 ml saline & 15 ml plain bupivacaine 0.25% Plus 150 units of hyaluronidase which is equal 1 ml ) .
  Interventions: Procedure: Ultrasound guided erector spinae plane block

INTERVENTIONS:
Procedure: Ultrasound guided erector spinae plane block — ESP block is most often performed using an in-plane ultrasound-guided technique. It is a paraspinal fascial plane block in which the needle placement is between the erector spinae muscle and the thoracic transverse processes, and a local anesthetic is administered, blocking the dorsal and ventral rami of the thoracic and abdominal spinal nerves

SUMMARY:
Evaluation of the postoperative pain via numeric rating scale (NRS) through erector spinae plane block (ESPB) by adding hyaluronidase as an adjuvant to bupivacaine on the postoperative analgesia in erector spinae plane block.

DETAILED DESCRIPTION:
* During mask preoxygenation, patients baseline hemodynamic parameters will be recorded regarding blood pressure and heart rate.
* General anesthesia will be standardized for all patients with :

  2 µg / kg fentanyl, 2 mg/kg 2% propofol then 0.5 mg/kg atracuriam will be administered for muscle relaxation.
* Patients will be intubated and lungs mechanically ventilated to maintain end-tidal CO2 between 30 to 35 mmHg. Fresh gas flow oxygen in air 30-40% at a rate of 3 L/min .
* The patients will receive 1.2 % MAC of isoflurane .
* Top- up doses of 0.15 mg/kg atracurium will be given to maintain intraoperative muscle relaxation.
* In all patients , insufflation will be under pressure of 15 mmHg or less .
* The surgical time in all surgical procedures will be fixed in the range of two hours and by the same surgical team.

After the patient will be generally anesthesized and before starting the operation , the erector spinae plane block will be performed .

• Patients will be randomly allocated to one of the two groups and the study will be double blinded where neither the operator nor the patients know which group will be . The syringes will be prepared by the other investigators.

. In group l : ESPB with bupivacaine 0.25% (30 ml volume : 15 ml saline Plus 15 ml plain bupivacaine ) .

In group ll : ESPB with plain bupivacaine 0.25% and hyaluronidase ( 14 ml saline & 15 ml plain bupivacaine 0.25% Plus 150 units of hyaluronidase which is equal 1 ml ) .

ESP block is most often performed using an in-plane ultrasound-guided technique. It is a paraspinal fascial plane block in which the needle placement is between the erector spinae muscle and the thoracic transverse processes, and a local anesthetic is administered, blocking the dorsal and ventral rami of the thoracic and abdominal spinal nerves (4).

USG-ESPB will be performed with the patient is in lateral position,The curvilinear ultrasound transducer should be placed in a cephalocaudal orientation over the midline of the back at the desired level. The probe should then slowly be moved laterally until the transverse process is visible. The transverse process requires differentiation from the rib at that level. The transverse process will be more superficial and wider, while the rib will be deeper and thinner. Upon verification of the transverse process, the trapezius muscle, rhomboid major muscle (if performing at T5 level or higher), and erector spinae muscle should be identified superficial to the transverse process. The Tuohy needle should be inserted superior to the ultrasound probe using an in-plane approach in the cephalad to caudal direction. The bevel of the Tuohy needle should point posteriorly and inferiorly, and advance under ultrasound guidance through the trapezius muscle, rhomboid major muscle, and erector spinae muscle and towards the transverse process; once the needle tip is below the erector spinae muscle, a small bolus of local anesthetic should be given through the Tuohy needle. The erector spinae muscle should be visualized, separating from the transverse process. This separation from the transverse process confirms the proper needle position. The local anesthetic should then be injected in 5 ml increments, with aspiration after every 5 ml to prevent intravascular injection.

* It is important to visualize the pleura very clearly at all times. The hyperechoic line of the pleura and underlying hyperechoic air artifacts move with respiration.
* Dose of hyaluronidase :

The minimum and maximum effective doses of hyaluronidase are unknown. The doses used range from 0.75 IU/mL to 300 IU/m.(8) (Table 3)

ELIGIBILITY:
Inclusion Criteria:

1. Elective percutaneous nephrolithotomy
2. Age: adult patients between 20 - 65 years old.
3. Gender: Both male and female.
4. ASA Class: I and II.

Exclusion Criteria:

1. Refusal of patient.
2. Patients ASA class III and IV.
3. Chronic kidney disease grade lll & lV .
4. Pregnancy and lactation.
5. Allergy to any of the study medications.
6. Addicts and drug abusers.
7. Patients taking corticosteroids or any cardio - active drugs.
8. Severe coagulopathy ( INR >3 or platelets <70*10) .
9. Fever or sepsis.
10. Local infection at site of the injection.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score by numeric rating scale (NRS) | Started measuring on admission to PACU ( 0 time) and 2, 4, 6 and 24 hours following admission
  Pain intensity will be estimated by a numeric rating scale (NRS) (0 = no pain, 10 = worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospitals, Cairo, Cairo Governorate, Egypt